CLINICAL TRIAL: NCT00773084
Title: Aliskiren and Renin Inhibition in Diastolic Heart Failure in Mexican Americans
Brief Title: Aliskiren and Renin Inhibition in Diastolic Heart Failure
Acronym: ARID-HF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in recruiting patients and then the PI left the institution
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Selim Krim, MD, Texas Tech University Health Sciences Center--Dept. of Internal Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARID-HF
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2011-03

CONDITIONS: Diastolic Heart Failure
Keywords: Diastolic Heart Failure; Hispanic Americans; Aliskiren; Spironolactone; Lisinopril; Diastolic Heart Failure in Hispanic Americans
MeSH Terms: conditions — Heart Failure, Diastolic | interventions — aliskiren; Spironolactone; Lisinopril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Drug (Active Comparator): Aliskiren plus spironolactone vs. Lisinopril plus spironolactone
  Interventions: Drug: Aliskiren plus spironolactone vs. Lisinopril plus spironolactone

INTERVENTIONS:
Drug: Aliskiren plus spironolactone vs. Lisinopril plus spironolactone — Subjects will be in the study for a total of 8 weeks. Subjects with stable diastolic HF on current ACEI therapy will be randomized into two treatment groups. The study group will receive Aliskiren plus spironolactone and the control group will receive Lisinopril plus spironolactone. These 2 groups will be further divided according to ethnicity: Mexican Americans and non-Hispanic whites. Sixty patients will be recruited, 30 per treatment group. Subjects will have a 2 week wash-out period. At the end of this period, blood will be collected and subjects will be asked to take the assigned medication once daily for 6 weeks. Subjects will be asked to return every 2 weeks at which time blood pressure, serum potassium and creatinine levels will be assessed. Their medications will be titrated depending on clinical tolerance and symptom control. At the end of 6 weeks of treatment blood markers will be drawn and differences will be analyzed.
  Other Names: Tekturna; Lisinopril; Spironolactone

SUMMARY:
This study is being conducted to compare the effects that 2 different combinations of heart failure medications have on the levels of certain blood markers which cause and/or worsen heart failure. Additionally, the investigators will investigate any differences that may exist between Hispanics and Non-Hispanics. The investigators hope to find that Hispanic Americans will have a greater response to this new regimen compared to non-Hispanic Americans.

DETAILED DESCRIPTION:
Our main hypothesis is that in contrast to non Hispanic whites, the degree of RAAS system activation is more pronounced in Mexican Americans with diastolic HF and consequently their response to RAAS inhibition therapy is greater. Blocking the RAAS with renin inhibitor plus aldosterone receptor blocker should produce measurable changes in biomarkers as well as physiologic improvement that could therefore translate into improved clinical outcomes. These changes should be greater appreciated in Mexican Americans if the central pathophysiologic influence of HF in this population was RAAS maladaptation.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic stable diastolic HF documented by clinical diagnosis and echocardiogram within the last 2 years
2. NYHA classes I-III, symptomatically stable (for >1month)
3. Age 21-70 years
4. Either of Hispanic ethnicity (Mexican American origin) or non-Hispanic white
5. Patients on ACE inhibitor therapy (lisinopril)
6. Blood pressure >100/75 mmHg
7. Adequate birth control
8. Patients seen in TTUHSC Cardiology or Internal Medicine clinic for at least two visits since January 2008

Exclusion Criteria:

1. Acute coronary syndrome (within the last month).
2. Recent acute diastolic or systolic HF (within the last month)
3. Pancreatic disease
4. Renal artery stenosis
5. Pregnancy
6. History of angioedema
7. Severe hypotension (systolic BP<90mmHg or mean arterial pressure <65mmHg)
8. Hyperkalemia (defined by K+>5 mEq/L)
9. Chronic Kidney Disease (Stage 3 and above)
10. Systolic dysfunction (ejection fraction below 50%)
11. Ethnicity other than Mexican American or non-Hispanic white

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-09; Primary Completion 2009-08 (Estimated); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
Compare the baseline level of RAAS dysregulation between Mexican Americans and non-Hispanic whites with stable diastolic HF by measuring established biomarkers. | 8 weeks
Evaluate the superiority of aliskiren plus spironolactone combination over an lisinopril plus spironolactone combination in inhibiting the RAAS system among patients with diastolic HF. | 8 weeks
Compare the clinical and biological benefit of RAAS system inhibition between aliskiren plus spironolactone and lisinopril plus spironolactone as measured by clinical indicators and serum biomarkers | 8 weeks
Assess ethnicity-specific differences in the clinical response to either RAAS inhibition treatment between Mexican Americans and non-Hispanic whites. | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Tech University Health Sciences Center, Lubbock, Texas, United States